CLINICAL TRIAL: NCT06709820
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY4060874 in Healthy Participants
Brief Title: A Study of LY4060874 in Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27300; J5X-MC-YJAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- LY4060874 (Part A Subcutaneous) (Experimental): Single ascending dose of LY4060874 administered subcutaneously (SC).
  Interventions: Drug: LY4060874
- LY4060874 (Part A Intravenous) (Experimental): Single ascending dose of LY4060874 administered intravenously (IV).
  Interventions: Drug: LY4060874
- LY4060874 (Part B) (Experimental): Multiple ascending doses of LY4060874 administered SC.
  Interventions: Drug: LY4060874
- LY4060874 (Part B Chinese) (Experimental): Multiple ascending doses of LY4060874 administered SC in Chinese participants.
  Interventions: Drug: LY4060874
- LY4060874 (Part C Japanese) (Experimental): Multiple ascending doses of LY4060874 administered SC in Japanese participants.
  Interventions: Drug: LY4060874
- Placebo (SC) (Placebo Comparator): Placebo administered SC in Part A, B, and C.
  Interventions: Drug: Placebo
- Placebo (IV) (Placebo Comparator): Placebo administered IV in Part A.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY4060874 — Administered SC
  Arms: LY4060874 (Part A Subcutaneous); LY4060874 (Part B Chinese); LY4060874 (Part B); LY4060874 (Part C Japanese)
Drug: LY4060874 — Administered IV
  Arms: LY4060874 (Part A Intravenous)
Drug: Placebo — Administered SC
  Arms: Placebo (SC)
Drug: Placebo — Administered IV
  Arms: Placebo (IV)

SUMMARY:
The purpose of this study is to evaluate safety and tolerability of LY4060874 in healthy participants.

Study participation may last up to 22 weeks and up to approximately 18 study visits.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation, including medical history and physical examination.
* Have a body mass index in the range of 20 to 29.9 kilogram per meter squared (kg/m²), inclusive, at screening.
* To qualify as Chinese for this study, all 4 of the participant's biological grandparents must be of exclusive Chinese descent and born in China.
* To qualify as a participant of first-generation Japanese origin, the participant, the participant's biological parents, and all the participants' biological grandparents must be of exclusive Japanese descent and born in Japan.

Exclusion Criteria:

* Have a history of or have been diagnosed with Type 1 or Type 2 diabetes mellitus.
* Have hemoglobin A1c (HbA1c) > 6.4% or 46 millimoles/mole (mmol/mol) at screening.
* Have taken approved, including over the counter (OTC) or prescribed, medication or investigational medication for weight loss, including GLP-1 receptor agonists, within the previous 3 months of study screening.
* Have had surgical treatment for obesity.
* Are actively participating in a weight loss program or intend to initiate an intensive diet and/or exercise program during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Baseline up to 22 Weeks
  Number of participants with one or more TEAEs and SAEs.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time (AUC) of LY4060874 | PK: Part A: Baseline up to 13 weeks; Part B and C: Baseline up to 18 weeks
  PK: Area Under the Concentration Versus Time (AUC) of LY4060874
PK: Maximum Observed Concentration of LY4060874 | PK: Part A: Baseline up to 13 weeks; Part B and C: Baseline up to 18 weeks
  PK: Cmax of LY4060874

CONTACTS AND LOCATIONS:
Overall Officials: 1-877-CTLILLY (1-877-285-4559) or 3176154559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Fortrea, Inc., Dallas, Texas, United States
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No